CLINICAL TRIAL: NCT02876913
Title: Evaluation on the Proper Size of the Nasotracheal Tube and Depth in Nasotracheal Intubation: a Preliminary Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2016-0504
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group Nasotracheal Intubation: Patients who are scheduled for nasotracheal intubation for general anesthesia

SUMMARY:
The nasotracheal intubation is preferred for oral surgery; it provides an easier view of the surgical field. However, nasotracheal tubes are produced by foreign countries. Tubes are often not fitted in anatomy of Korean people because of small nostril. When the size of the tube is chosen by nostril size, the length of nasotracheal tube is not appropriate to the glottis. The aim of this study is to evaluate on the proper size of the nasotracheal tube and depth in nasotracheal intubation in Korean. Forty patients (20 males and 20 females) who are scheduled for nasal intubation for general anesthesia will be enrolled. The primary outcome is the proportion of patients who are in inappropriate insertion of nasotracheal tube; the proximal end of tube's cuff is less than 2 cm below vocal cord. The size of nostril, length from the nare to the carina and vocal cord are measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for nasotracheal intubation for general anesthesia

Exclusion Criteria:

* age < 20 years and age > 70 years
* ASA(American Society of Anesthesiologist) class III or more
* pregnancy
* emergency surgery
* nasal airway disease
* expected difficult intubation (difficult intubation history, Modified Mallampati score 4, mouth opening <2cm, facial anomaly)
* unstable teeth

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for nasotracheal intubation for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Proportion of the inappropriate insertion of nasotracheal tube | 5 minutes after induction of general anesthesia
  the inappropriate insertion of nasotracheal tube; the proximal end of tube's cuff is less than 2 cm below vocal cord

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee B, Park WK, Yun SY, Kang S, Kim HJ. Insertion depth of nasotracheal tubes sized to fit the nostril: an observational study. J Int Med Res. 2019 Jan;47(1):235-243. doi: 10.1177/0300060518800105. Epub 2018 Dec 16. PMID 30556457